CLINICAL TRIAL: NCT03512275
Title: A Phase II, Open Label Study of Bermekimab in Patients With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study of Bermekimab in Patients With Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-PT045
Record Dates: First submitted 2018-04-11; First posted 2018-04-30 (Actual); Results first posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 400mg cohort, no prior treatment with anti-TNF agent(s) (Experimental): N=10 patients that have had no prior treatment with biological agents that block TNF will receive a total of 13 X 400mg subcutaneous injections of bermekimab. Dosing will occur weekly for 12 weeks, inclusive of visit 1 and visit 13.
  Interventions: Drug: Bermekimab Monoclonal Antibody 400 mg
- 400 mg cohort, prior treatment with anti-TNF agent(s) (Experimental): N=10 patients that have failed anti-TNF therapy will receive a total of 13 X 400mg subcutaneous injections of bermekimab. Dosing will occur weekly for 12 weeks, inclusive of visit 1 and visit 13.
  Interventions: Drug: Bermekimab Monoclonal Antibody 400 mg

INTERVENTIONS:
Drug: Bermekimab Monoclonal Antibody 400 mg — subcutaneous injection
  Other Names: MABp1

SUMMARY:
Phase 2 study of bermekimab in patients with moderate to severe Hidradenitis Suppurativa.

DETAILED DESCRIPTION:
Phase 2, open label study of bermekimab in patients with moderate to severe Hidradenitis Suppurativa. The study is multicenter and will consist of two patient groups, each of which will receive a total of 13 X 400mg weekly subcutaneous injections of bermekimab: Group A (n=10) patients who have failed anti-TNF therapy, and Group B (n=10) patients who have had no prior treatment with biological agents that block TNF.

Patients will be followed for 13 weeks to allow for assessment of safety and preliminary efficacy.

Additionally, patients who had received the 200 mg weekly subcutaneous injections of bermekimab under the previous version of this protocol are eligible to begin receiving the 400 mg dose starting with his/her next scheduled visit, and for the remainder of his/her treatment plan.

XBiotech owned bermekimab and sponsored and completed study prior to Dec 30, 2019.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided by the patient.
* Male or female, age 18 years or greater.
* For group A, patients must have received and failed anti-TNF therapy.

  * For Group B, patients must not have received any prior treatment with any anti-TNF therapy.
  * Patients who have received 200 mg dose of bermekimab in this study (previous version(s)) are eligible to begin receiving 400 mg dose starting with the patient's next scheduled visit for the remainder of his/her treatment plan.
* Diagnosis of HS for at least 1 year prior to screening.
* HS affecting at least two distinct anatomic areas, one of which is Hurley II or III stage.
* A total body count of abscesses and inflammatory nodules (AN) of at least 3
* Full understanding of the procedures of the study protocol and willingness to comply with them.
* In case of female patients of childbearing potential, willingness to use one method of contraception of high efficacy during the entire study period. This method can be intake of hormonal contraceptives or the use of one of the following: condoms, diaphragm or an intrauterine device. Women of non-childbearing potential include those considered to have a medical history that indicates that pregnancy is not a reasonable risk, including post-menopausal women and those with a history of hysterectomy.

Exclusion Criteria:

* Age below 18 years.
* Receipt of oral antibiotic treatment for HS within 28 days prior to screening.
* Receipt of prescription topical therapies for the treatment of HS within 14 days prior to screening, and/or systemic therapies for HS (immunosuppressants, corticosteroids, retinoids, or hormonal therapies) within 28 days prior to screening.
* History of treatment with bermekimab for any reason, EXCEPT patients previously treated with 200 mg bermekimab dose in the previous version(s) of this study.
* History of severe allergic or anaphylactic reactions to human, humanized, chimeric, or murine monoclonal antibodies.
* Has received a live (attenuated) vaccine over the 4 weeks prior to screening.
* New intake of opioid analgesics starting within 14 days prior to screening.
* Major surgery (requiring general anesthesia or respiratory assistance) within 28 days prior to Visit 1, Day 0 of start of study drug.
* Hepatic dysfunction defined as any value of transaminases or of γ-glutamyl transpeptidase (γGT), or of total bilirubin > 3 x upper normal limit
* Stage C Child-Pugh liver cirrhosis.
* Chronic infection by the human immunodeficiency virus (HIV), hepatitis B virus (HBV) and/or hepatitis C virus (HCV).
* Neutropenia defined as <1,000 neutrophils/mm3.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tennessee Clinical Research Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: CSR
Time Frame: Starting from time of study completion and for the next year
Access Criteria: The Clinical Study Report (CSR) will be distributed to clinical sites who participated in the study.

REFERENCES:
- [Derived] Gottlieb A, Natsis NE, Kerdel F, Forman S, Gonzalez E, Jimenez G, Hernandez L, Kaffenberger J, Guido G, Lucas K, Montes D, Gold M, Babcock C, Simard J. A Phase II Open-Label Study of Bermekimab in Patients with Hidradenitis Suppurativa Shows Resolution of Inflammatory Lesions and Pain. J Invest Dermatol. 2020 Aug;140(8):1538-1545.e2. doi: 10.1016/j.jid.2019.10.024. Epub 2020 Jan 29. PMID 32004568

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed): Participants who did not respond to anti-TNF therapy, received bermekimab subcutaneously at a dose of 400 mg weekly (13 doses). Participants were followed for 13 weeks to allow for assessment of safety and preliminary efficacy.
- Group B: Bermekimab 400 mg (Anti-TNF Naive): Participants who did not receive prior treatment with biological agents that block TNF received bermekimab subcutaneously at a dose of 400 mg weekly (13 doses). Participants were followed for 13 weeks to allow for assessment of safety and preliminary efficacy.
Period: Overall Study
Arm/Group | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) | Group B: Bermekimab 400 mg (Anti-TNF Naive)
Started | 24 | 18
Completed | 22 | 11
Not Completed | 2 | 7
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 3
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) | Group B: Bermekimab 400 mg (Anti-TNF Naive) | Total
Number analyzed (Participants) | 24 | 18 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 18 | 41
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (13.14) | 41.5 (12.02) | 39.8 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 9 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 18 | 15 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 24 | 18 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event is defined as any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical or biological agent under study.
Time Frame: Up to Visit 14 (up to Day 93)
Population: The safety analysis set (SAF) consisted of all participants that received at least one dose of study medication and were analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) | Group B: Bermekimab 400 mg (Anti-TNF Naive)
Number analyzed (Participants) | 24 | 18
Participants | 21 | 16

2. Secondary Outcome: Percentage of Participants Achieving Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 12
Description: Percentage of participants achieving HiSCR at Week 12 was reported. For this score participants were defined as achievers or non-achievers. The positive HiSCR score was defined as a greater than or equal to (>=) 50% reduction in inflammatory lesion AN count (sum of abscesses and inflammatory nodules), and no increase in abscesses or draining fistulas in hidradenitis suppurativa compared with the lesions counted on visit 1 (baseline).
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) | Group B: Bermekimab 400 mg (Anti-TNF Naive)
Number analyzed (Participants) | 24 | 18
Percentage of Participants | 62.5 | 61.1

3. Secondary Outcome: Plasma Concentration of Bermekimab
Description: An enzyme-linked immunosorbent assay (ELISA) was developed to specifically measure bermekimab levels in human plasma. The blood samples were collected at each pharmacokinetic (PK) collection time point for PK analysis.
Time Frame: Predose at Days 14 (Visit 3), 28 (Visit 5), 56 (Visit 9), 84 (Visit 13)
Population: The safety analysis set (SAF) consisted of all participants that received at least one dose of study medication and were analyzed as treated. Here, 'N' (number of participants analyzed) is defined as participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) | Group B: Bermekimab 400 mg (Anti-TNF Naive)
Number analyzed (Participants) | 23 | 16
micrograms per milliliter (mcg/mL)
  Visit 3 | 32.7 (18.3) | 36.7 (22.7)
  Visit 5 | 37.4 (20.7) | 42.2 (25.0)
  Visit 9 | 36.3 (20.9) | 48.0 (31.7)
  Visit 13 | 42.1 (21.1) | 55.8 (43.6)

4. Secondary Outcome: Change From Baseline to Week 12 in Visual Analog Scale (VAS) Score for Disease
Description: Change from baseline in VAS score for disease was reported. The VAS is a validated, subjective measure for participants disease impression. Disease impression scores were recorded using a similar scale, with 0 representing "not at all severe" and 10 representing "extremely severe".
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) | Group B: Bermekimab 400 mg (Anti-TNF Naive)
Number analyzed (Participants) | 24 | 18
Units on scale | 3.11 (0.61) | 3.71 (0.75)

5. Secondary Outcome: Change From Baseline to Week 12 in VAS Score for Pain
Description: Change from baseline in VAS score for pain was reported. The VAS is a validated, subjective measure for acute and chronic pain. Pain scores were recorded by marking a number on a scale from 0 to 10, 0 representing "no pain" and 10 representing "extremely painful".
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) | Group B: Bermekimab 400 mg (Anti-TNF Naive)
Number analyzed (Participants) | 24 | 18
Units on scale | 4.07 (0.64) | 5.01 (0.79)

6. Secondary Outcome: Change From Baseline to Week 12 in Dermatology Life Quality Index (DLQI) Score
Description: The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of disease symptoms and treatment on Quality of life (QOL). The format is a simple response (0 to 3 where 0 is "not at all" and 3 is "very much") to 10 questions, which assess QOL over the past week, with an overall scoring system of 0 to 30; a high score is indicative of a poor QOL.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) | Group B: Bermekimab 400 mg (Anti-TNF Naive)
Number analyzed (Participants) | 24 | 18
Units on scale | 7.03 (1.51) | 11.52 (1.85)

7. Secondary Outcome: Change From Baseline to Week 12 in Physician's Global Assessment (PGA) Score
Description: PGA is a physician's assessment of the severity of disease based on a 6-point scale (Clear [0], minimal [1], mild [2], moderate [3], severe [4], more severe [5]) ranging from 0-5. Higher score indicated more severity of disease.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) | Group B: Bermekimab 400 mg (Anti-TNF Naive)
Number analyzed (Participants) | 24 | 18
Units on scale | 0.81 (0.24) | 1.97 (0.30)

8. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS) at Week 12
Description: The DAS is the sum of scores of all affected areas of each participant. Each area was evaluated by the following formula: (the sum of the two largest diameters in each affected area in millimeter [mm]) * (Total number of lesions in the anatomic area multiplied by the degree of inflammation of each lesion on a scale of 0 to 3). A minimum score of 0 and there is no maximum score range. Higher scores indicate more disease activity.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) | Group B: Bermekimab 400 mg (Anti-TNF Naive)
Number analyzed (Participants) | 24 | 18
Units on scale | 35.56 (14.96) | 63.84 (18.35)

9. Secondary Outcome: Change From Baseline to Week 12 in Modified Sartorius Score (mSS)
Description: mSS is used to quantify severity of HS. Points are awarded for 12 body areas (left-right axillae, left - right sub/inframammary areas, intermammary area, left - right buttocks, left-right inguinocrural folds, perianal area, perineal area and other): points were awarded for nodules (2 points each);abscesses (4points);fistulas (4points);scars (1point); other findings (1 point); and longest distance between two lesions (no active lesion or only 1 lesion equal to [=]0 points, less than [<]5cm=2points, 5-10cm=4points, greater than [>]10cm 6points) and if lesions are separated by normal skin (yes-0 points; no-6points). Total mSS is sum of the 12 regional scores. Change from baseline in mSS was not reported as the electronic data capture (EDC) system erroneously requested data for this endpoint to be input in centimeters versus millimeters and conversion was not possible because it was given in ranges. Therefore, there was not enough valid data to sufficiently perform this endpoint analysis.
Time Frame: Baseline and Week 12
Population: The safety analysis set (SAF) consisted of all participants that received at least one dose of study medication and were analyzed as treated. Data was not collected and analyzed for this outcome measure due to change in planned analysis.
Arm/Group | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) | Group B: Bermekimab 400 mg (Anti-TNF Naive)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline to Week 12 in Inflammatory Lesion (Abscesses and Inflammatory Nodules) Count
Description: Change from baseline to Week 12 in inflammatory lesion (abscesses and inflammatory nodules) count was reported. The sum of abscesses and inflammatory nodules was measured for each participant to assess change in inflammatory lesion counts.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Count of lesions
Arm/Group | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) | Group B: Bermekimab 400 mg (Anti-TNF Naive)
Number analyzed (Participants) | 24 | 18
Count of lesions | 6.44 (1.03) | 3.97 (1.29)

11. Secondary Outcome: Change From Baseline to Week 12 in Hospital Anxiety Depression Scale (HADS)
Description: The HADS is an instrument for screening anxiety and depression in non-psychiatric populations; repeated administration also provides information about changes to a patient's emotional state. The HADS consisted of 14 items, 7 each for anxiety and depression symptoms; possible scores range from 0 to 21 for each subscale. The following cut-off scores were recommended for both subscales: 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety or depression.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) | Group B: Bermekimab 400 mg (Anti-TNF Naive)
Number analyzed (Participants) | 24 | 18
units on a scale
  HADS Anxiety Score | 3.11 (0.88) | 1.33 (1.08)
  HADS Depression Score | 1.39 (0.57) | 0.54 (0.70)

ADVERSE EVENTS:
Time Frame: Up to Visit 14 (up to Day 93)
Description: The safety analysis set (SAF) consists of all participants that receive at least one dose of study medication and will be analyzed as treated.
Arm/Group | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) | Group B: Bermekimab 400 mg (Anti-TNF Naive)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/18
Serious Adverse Events (participants affected / at risk) | 2/24 | 0/18
Other Adverse Events (participants affected / at risk) | 6/24 | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) (N=24) | Group B: Bermekimab 400 mg (Anti-TNF Naive) (N=18)
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Bermekimab 400 Milligram (mg) (Anti-Tumor Necrosis Factor [TNF] Failed) (N=24) | Group B: Bermekimab 400 mg (Anti-TNF Naive) (N=18)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Injection Site Erythema (General disorders) | 2 | 0
Injection Site Reaction (General disorders) | 2 | 2
Cellulitis (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Penile Oedema (Reproductive system and breast disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study will be published and/or presented at scientific meetings in a timely manner. The publication policy is described in the contract between the Sponsor and Investigator.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT03512275/Prot_SAP_001.pdf